CLINICAL TRIAL: NCT01663129
Title: Steroid-Induced Osteoporosis in the Pediatric Population - Canadian Incidence Study (STOPP-CIS)
Brief Title: Steroid-Induced Osteoporosis in the Pediatric Population - Canadian Incidence Study
Acronym: STOPP-CIS
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Leanne Ward, Director, Pediatric Bone Health Clinical and Research Programs, Children's Hospital of Eastern Ontario
Other Study IDs: 03-07e; 03-07e (Other: CHEO REB Protocol Number)
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Acute Lymphoblastic Leukemia; Nephrotic Syndrome; Rheumatism
Keywords: Children; Osteoporosis; Vertebral Compression Fractures; Chronic Illness; Glucocorticoids; Bone Fragility
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Nephrotic Syndrome; Rheumatic Diseases; Osteoporosis; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Leukemia Patient Group: Acute Lymphoblastic Leukemia (ALL)
- Rheumatic Disease Patient Group: * Juvenile Idiopathic Arthritis (JIA)
  * Systemic Lupus Erythematosis
  * Juvenile Dermatomyositis
  * Scleroderma
  * Overlap Syndromes
  * Sjogren's syndrome
  * Sarcoidosis
  * Systemic Vasculitis (excluding Kawasaki's disease and Henoch-Schonlein Purpura)
  * Systemic vasculitis as defined by the Chapel Hill Concensus Conference on Nomenclature. Other forms of systemic vasculitis, including Giant cell (temporal) arteritis, Takayasu's arteritis, Polyarteritis nodosa, Wegener's granulomatosis, Churg-Strauss syndrome, Microscopic polyangiitis, Essential cryoglobulinemic vasculitis, Cutaneous leukocytoclastic angiitis, Behcet's disease, Other vasculitis
  * Other rheumatic disease
- Nephrotic Syndrome Patient Group: Nephrotic syndrome will be classified according to the following categories:
  Idiopathic nephrotic syndrome, without renal biopsy histology, presumed minimal change disease (MCD), Focal segmental glomerulosclerosis (FSGS), confirmed on biopsy, Minimal change disease, confirmed on biopsy Nephrotic syndrome with Henoch-Schonlein Purpura (HSP).

SUMMARY:
To determine the magnitude and rate of bone mass deficits following initiation of glucocorticoid therapy for the treatment of pediatric leukemia, rheumatic conditions and nephrotic syndrome, we propose a 6 year, prospective study in 12 academic, tertiary care centres across Canada.

The investigators hypothesize that glucocorticoid-treated children with leukemia, rheumatic conditions and nephrotic syndrome will fail to accrue bone mass at a normal rate, and that deficits in mineral accrual will occur in a glucocorticoid dose- and duration-dependent fashion. We also hypothesize that the fracture incidence will increase with concomitant reductions in bone mass.

DETAILED DESCRIPTION:
Leukemia and Bone Morbidity Acute lymphoblastic leukemia (ALL) is the most common pediatric malignancy, with an overall survival rate now exceeding 70%. As such, there is an increasing population of survivors who are at risk for long-term sequelae of childhood leukemia, including osteoporosis. In Canada, there are approximately 250 new cases of childhood ALL diagnosed per year. All children in Canada undergoing therapy for the treatment of ALL in tertiary care pediatric hospitals will receive high dose glucocorticoids as per one of three ALL protocols (the Children's Cancer Group protocol, the Pediatric Oncology Group protocol, or the Dana Farber Cancer Institute Consortium protocol), depending upon the standard of care at a given institution. Musculoskeletal pain and gait abnormalities have been reported in one third of children with ALL at diagnosis, a sub-set of whom also demonstrate fractures. Radiographs of painful regions show metaphyseal lucencies, sclerotic lesions and sites of periosteal reaction in many of the patients with bone pain at presentation. Lumbar spine areal bone mineral density (BMD) is reduced at diagnosis, while total body and volumetric BMD are within the normal range. Several groups have reported significant loss of bone mass during therapy for ALL, while studies of bone mass restitution following chemotherapy have led to inconsistent results. The most rapid reductions in bone mass have occurred in the first 6-8 months of therapy, similar to the observed glucocorticoid effect on bone in adults. Fractures have been present in as many as 13% of children at diagnosis, rising to 39% during chemotherapy. In addition to glucocorticoids, a number of other mechanisms have been proposed for the skeletal morbidity in ALL, including infiltration of bone by leukemic cells, paraneoplastic factors, other medications, physical inactivity, cranial irradiation, inadequate nutrition and disordered mineral metabolism.

Rheumatic Conditions and Bone Morbidity Rheumatic diseases of childhood, including juvenile rheumatoid arthritis, systemic lupus erythematosis and juvenile dermatomyositis, are well-known to be associated with compromised skeletal health. Of these, juvenile rheumatoid arthritis has been evaluated the most extensively. Significant reductions in bone mass have been documented in a number of studies of pediatric patients with chronic rheumatic disease, and atraumatic fractures have been noted at an early age. Active arthritis may affect bone metabolism in areas adjacent to affected joints ("periarticular osteopenia"), and at more distant sites including the radius, spine, and femoral neck. In a recent study of pediatric patients with reductions in bone mass secondary to chronic rheumatic disease, 8/38 (21%) of patients had fragility fractures, primarily of the vertebrae. Similar to other osteoporotic conditions due to chronic illness, the pathogenesis of the bone morbidity in these cases is multi-factorial, with disease activity, muscle disease, physical inactivity, nutritional status and medical therapy playing significant roles. However, as in leukemia, glucocorticoid use has emerged as one of the strongest determinants of skeletal morbidity during treatment for juvenile rheumatoid arthritis and systemic lupus erythematosis. The role of glucocorticoids in bone morbidity associated with pediatric rheumatic diseases such as juvenile dermatomyositis and vasculitides has not been determined.

Nephrotic Syndrome and Bone Morbidity Childhood nephrotic syndrome is an idiopathic disorder characterized by proteinuria, hypoproteinemia, edema and hyperlipidemia. The incidence of the syndrome varies between 1:15,000 to 1:50,000. Following the introduction of glucocorticoid therapy in the 1970's, the mortality from nephrotic syndrome decreased dramatically over the ensuing 15 years, from 35 to 3 per cent. The vast majority of patients with nephrotic syndrome have steroid-responsive disease. In Canada, the standard of care for children with their first episode of nephrotic syndrome is high-dose glucocorticoid therapy for 6 weeks, followed by gradual tapering over the next three to seven months. Only one-third of patients will enter into permanent remission with this regime, while another third will require pulse steroid therapy for up to six weeks' duration at infrequent intervals throughout the growing years. The final third of patients will either require frequent courses of pulse glucocorticoid therapy or chronic steroid administration in order to achieve remission. Children with nephrotic syndrome are typically well-nourished, fully ambulatory, and otherwise well between episodes. Furthermore, their treatment regime is more likely to be characterized by glucocorticoid therapy alone, compared to the polytherapy that is required for the treatment of leukemia and rheumatic conditions. As such, the greater homogeneity of the nephrotic syndrome population allows for a more "pure" assessment of glucocorticoid effect on pediatric bone. Small studies have demonstrated reductions in bone mass by dual energy x-ray absorptiometry (DXA) and an increase in biochemical markers of bone resorption among young, glucocorticoid-treated patients with nephrotic syndrome. Tenbrock et al. recently showed by peripheral quantitative computed tomography that 16 children with nephrotic syndrome, all previously treated with glucocorticoids, had reductions in cortical area at the distal radius, which correlated with reductions in grip strength. The fracture rate among children with nephrotic syndrome is presently unknown. Among adults with nephrotic syndrome, high-dose glucocorticoid administration led to rapid bone loss in the first few months of therapy, raising the question whether preventive therapy should be initiated in such adults after three months of glucocorticoid use, if measures of bone mass have fallen significantly below baseline.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Children aged > or = 1 month to < or = 16 years at the time of enrolment.
2. Clinical diagnosis of one of the following three diseases:

   1. Acute lymphoblastic leukemia OR
   2. Rheumatic disease,OR
   3. Nephrotic syndrome
3. Need for the first-time initiation of intravenous (IV) or oral glucocorticoid therapy (regardless of the dose or duration) for the treatment of the leukemia, nephrotic syndrome or rheumatic conditions, as determined by the attending physician. IV and oral glucocorticoids used in current clinical practice for the treatment of leukemia, nephrotic syndrome and rheumatic conditions include cortisone, hydrocortisone, methylprednisolone, prednisolone, prednisone, dexamethasone, and deflazacorte. If patients are receiving intra-articular, inhaled, intra-nasal or topical corticosteroids, these agents alone do not meet the steroid criteria for enrolment in the study. However, the use of such steroids will be captured as part of the Case Report Form.
4. Only patients who are receiving glucocorticoids for the first time for the treatment of their underlying leukemia, nephrotic syndrome or rheumatic condition, will be included. Patients who have received glucocorticoids in the past for other indications (e.g. asthma), may be included in the study, provided they have not received more than 14 consecutive days of IV or oral steroids in the 12 months prior to the first initiation of steroids for their underlying leukemia, nephrotic syndrome or rheumatic condition. The pre-STOPP study use of glucocorticoids for 14 days or less, for treatment of unrelated medical conditions in the 12 months prior to the first initiation of steroids to treat the underlying leukemia, nephrotic syndrome or rheumatic conditions, will be captured in the Case Report Form.
5. Informed consent.
6. Ability and willingness to maintain a "Glucocorticoid Dose Diary" throughout the study.
7. For menstruating females, a negative pregnancy test will be required prior to enrolment.

Exclusion Criteria:

1. Inability to obtain baseline investigations within 30 days of the first-time initiation of glucocorticoids for the treatment of the underlying leukemia, nephrotic syndrome or rheumatic condition.
2. Complete immobilization (patient confined to bed except for toileting) for more than 14 consecutive days in the 12 months prior to the initiation of glucocorticoids for the treatment of their underlying leukemia, nephrotic syndrome or rheumatic condition.
3. Use of IV or oral glucocorticoids for more than 14 consecutive days, for the treatment of unrelated medical conditions, in the 12 months prior to the first initiation of steroids for the treatment of the underlying leukemia, nephrotic syndrome or rheumatic condition.
4. Treatment of osteoporosis with medical therapy prior to the initial baseline visit (treatment with, for example, a bisphosphonate, calcitonin, fluoride).
5. Unwillingness to utilize a medically approved method of birth control if menstruating and sexually active.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be recruited into the study following a clinical diagnosis of glucocorticoid-requiring leukemia, rheumatic disease or nephrotic syndrome, as determined by the study collaborators in each of the three sub-specialties according to their usual clinical practice. Potential participants will be identified by the attending physician (oncologist, rheumatologist or nephrologist) who will then refer the patient to the site bone designee. The bone designee (or his/her research assistant) will be responsible for determining patient eligibility and for carrying out the requirements of the study.
Sampling Method: Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2005-01; Primary Completion 2014-03-06 (Actual); Study Completion 2014-03-06 (Actual)

PRIMARY OUTCOMES:
The magnitude and rate of total body, hip and lumbar spine bone mass deficits | up to 72 months (plus at 3 months post baseline visit for the Nephrotic Syndrome Group)
  We will determine the magnitude and rate of total body, hip and lumbar spine bone mass deficits following initiation of glucocorticoid therapy, in relation to glucocorticoid dose and duration, among children with leukemia, rheumatic conditions and nephrotic syndrome. The longitudinal pattern of deficits (or gains) in bone mass will be determined for each disease state by plotting bone mass measurements taken at 6 month intervals throughout the study, with an additional 3 month measurement being recorded for patients with nephrotic syndrome.

SECONDARY OUTCOMES:
Glucocorticoid threshold dose | At baseline, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66 and 72-month visits
  To identify whether a glucocorticoid threshold dose exists for each of the three disease categories, above which significant deficits in bone mass are likely to occur.
Frequency of atraumatic fractures | At baseline, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66 and 72-month visits
  To assess the frequency of atraumatic fractures in relation to glucocorticoid dose and duration for each of the three chronic illnesses.
Fracture risk | At baseline, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66 and 72-month visits
  To determine the fracture risk associated with a given reduction in bone mass from baseline, for each of the three chronic diseases.
Magnitude of bone mass restitution | At baseline, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66 and 72-month visits
  To determine the magnitude of bone mass restitution when glucocorticoid therapy is withdrawn, and to evaluate whether recovery is age- and/or pubertal stage-dependent.
Handedness and lateralization of bone density | Once during either the baseline, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66 or 72-month visits
  To investigate the relationship between handedness and lateralization of bone density.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Ward, MD FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (12):
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Winnipeg Children's Hospital, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Shriners Hospital for Children, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Feber J, Gaboury I, Ni A, Alos N, Arora S, Bell L, Blydt-Hansen T, Clarson C, Filler G, Hay J, Hebert D, Lentle B, Matzinger M, Midgley J, Moher D, Pinsk M, Rauch F, Rodd C, Shenouda N, Siminoski K, Ward LM; Canadian STOPP Consortium. Skeletal findings in children recently initiating glucocorticoids for the treatment of nephrotic syndrome. Osteoporos Int. 2012 Feb;23(2):751-60. doi: 10.1007/s00198-011-1621-2. Epub 2011 Apr 15. PMID 21494860
- [Result] Huber AM, Gaboury I, Cabral DA, Lang B, Ni A, Stephure D, Taback S, Dent P, Ellsworth J, LeBlanc C, Saint-Cyr C, Scuccimarri R, Hay J, Lentle B, Matzinger M, Shenouda N, Moher D, Rauch F, Siminoski K, Ward LM; Canadian Steroid-Associated Osteoporosis in the Pediatric Population (STOPP) Consortium. Prevalent vertebral fractures among children initiating glucocorticoid therapy for the treatment of rheumatic disorders. Arthritis Care Res (Hoboken). 2010 Apr;62(4):516-26. doi: 10.1002/acr.20171. PMID 20391507
- [Result] Halton J, Gaboury I, Grant R, Alos N, Cummings EA, Matzinger M, Shenouda N, Lentle B, Abish S, Atkinson S, Cairney E, Dix D, Israels S, Stephure D, Wilson B, Hay J, Moher D, Rauch F, Siminoski K, Ward LM; Canadian STOPP Consortium. Advanced vertebral fracture among newly diagnosed children with acute lymphoblastic leukemia: results of the Canadian Steroid-Associated Osteoporosis in the Pediatric Population (STOPP) research program. J Bone Miner Res. 2009 Jul;24(7):1326-34. doi: 10.1359/jbmr.090202. PMID 19210218
- [Result] Rodd C, Lang B, Ramsay T, Alos N, Huber AM, Cabral DA, Scuccimarri R, Miettunen PM, Roth J, Atkinson SA, Couch R, Cummings EA, Dent PB, Ellsworth J, Hay J, Houghton K, Jurencak R, Larche M, LeBlanc C, Oen K, Saint-Cyr C, Stein R, Stephure D, Taback S, Lentle B, Matzinger M, Shenouda N, Moher D, Rauch F, Siminoski K, Ward LM; Canadian Steroid-Associated Osteoporosis in the Pediatric Population (STOPP) Consortium. Incident vertebral fractures among children with rheumatic disorders 12 months after glucocorticoid initiation: a national observational study. Arthritis Care Res (Hoboken). 2012 Jan;64(1):122-31. doi: 10.1002/acr.20589. PMID 22213727
- [Result] Alos N, Grant RM, Ramsay T, Halton J, Cummings EA, Miettunen PM, Abish S, Atkinson S, Barr R, Cabral DA, Cairney E, Couch R, Dix DB, Fernandez CV, Hay J, Israels S, Laverdiere C, Lentle B, Lewis V, Matzinger M, Rodd C, Shenouda N, Stein R, Stephure D, Taback S, Wilson B, Williams K, Rauch F, Siminoski K, Ward LM. High incidence of vertebral fractures in children with acute lymphoblastic leukemia 12 months after the initiation of therapy. J Clin Oncol. 2012 Aug 1;30(22):2760-7. doi: 10.1200/JCO.2011.40.4830. Epub 2012 Jun 25. PMID 22734031
- [Result] Siminoski K, Lee KC, Jen H, Warshawski R, Matzinger MA, Shenouda N, Charron M, Coblentz C, Dubois J, Kloiber R, Nadel H, O'Brien K, Reed M, Sparrow K, Webber C, Lentle B, Ward LM; STOPP Consortium. Anatomical distribution of vertebral fractures: comparison of pediatric and adult spines. Osteoporos Int. 2012 Jul;23(7):1999-2008. doi: 10.1007/s00198-011-1837-1. Epub 2011 Nov 23. PMID 22109742
- [Result] Siminoski K, Lee KC, Abish S, Alos N, Bell L, Blydt-Hansen T, Couch R, Cummings EA, Ellsworth J, Feber J, Fernandez CV, Halton J, Huber AM, Israels S, Jurencak R, Lang B, Laverdiere C, LeBlanc C, Lewis V, Midgley J, Miettunen PM, Oen K, Phan V, Pinsk M, Rauch F, Rodd C, Roth J, Saint-Cyr C, Scuccimarri R, Stephure D, Taback S, Wilson B, Ward LM; Canadian STOPP Consortium National Pediatric Bone Health Working Group. The development of bone mineral lateralization in the arms. Osteoporos Int. 2013 Mar;24(3):999-1006. doi: 10.1007/s00198-012-2054-2. Epub 2012 Jun 29. PMID 22744715
- [Result] Cummings EA, Ma J, Fernandez CV, Halton J, Alos N, Miettunen PM, Jaremko JL, Ho J, Shenouda N, Matzinger MA, Lentle B, Stephure D, Stein R, Sbrocchi AM, Rodd C, Lang B, Israels S, Grant RM, Couch R, Barr R, Hay J, Rauch F, Siminoski K, Ward LM; Canadian STOPP Consortium (National Pediatric Bone Health Working Group). Incident Vertebral Fractures in Children With Leukemia During the Four Years Following Diagnosis. J Clin Endocrinol Metab. 2015 Sep;100(9):3408-17. doi: 10.1210/JC.2015-2176. Epub 2015 Jul 14. PMID 26171800
- [Result] Ward LM, Ma J, Lang B, Ho J, Alos N, Matzinger MA, Shenouda N, Lentle B, Jaremko JL, Wilson B, Stephure D, Stein R, Sbrocchi AM, Rodd C, Lewis V, Israels S, Grant RM, Fernandez CV, Dix DB, Cummings EA, Couch R, Cairney E, Barr R, Abish S, Atkinson SA, Hay J, Rauch F, Moher D, Siminoski K, Halton J; Steroid-Associated Osteoporosis in the Pediatric Population (STOPP) Consortium. Bone Morbidity and Recovery in Children With Acute Lymphoblastic Leukemia: Results of a Six-Year Prospective Cohort Study. J Bone Miner Res. 2018 Aug;33(8):1435-1443. doi: 10.1002/jbmr.3447. Epub 2018 May 22. PMID 29786884
- [Result] LeBlanc CM, Ma J, Taljaard M, Roth J, Scuccimarri R, Miettunen P, Lang B, Huber AM, Houghton K, Jaremko JL, Ho J, Shenouda N, Matzinger MA, Lentle B, Stein R, Sbrocchi AM, Oen K, Rodd C, Jurencak R, Cummings EA, Couch R, Cabral DA, Atkinson S, Alos N, Rauch F, Siminoski K, Ward LM; Canadian STeroid-Associated Osteoporosis in Pediatric Population (STOPP) Consortium. Incident Vertebral Fractures and Risk Factors in the First Three Years Following Glucocorticoid Initiation Among Pediatric Patients With Rheumatic Disorders. J Bone Miner Res. 2015 Sep;30(9):1667-75. doi: 10.1002/jbmr.2511. Epub 2015 May 26. PMID 25801315
- [Result] Ma J, Siminoski K, Alos N, Halton J, Ho J, Lentle B, Matzinger M, Shenouda N, Atkinson S, Barr R, Cabral DA, Couch R, Cummings EA, Fernandez CV, Grant RM, Rodd C, Sbrocchi AM, Scharke M, Rauch F, Ward LM; Canadian STOPP Consortium. The choice of normative pediatric reference database changes spine bone mineral density Z-scores but not the relationship between bone mineral density and prevalent vertebral fractures. J Clin Endocrinol Metab. 2015 Mar;100(3):1018-27. doi: 10.1210/jc.2014-3096. Epub 2014 Dec 11. PMID 25494661
- [Result] Jaremko JL, Siminoski K, Firth GB, Matzinger MA, Shenouda N, Konji VN, Roth J, Sbrocchi AM, Reed MH, O'Brien MK, Nadel H, McKillop S, Kloiber R, Dubois J, Coblentz C, Charron M, Ward LM; Canadian STOPP Consortium National Pediatric Bone Health Working Group. Common normal variants of pediatric vertebral development that mimic fractures: a pictorial review from a national longitudinal bone health study. Pediatr Radiol. 2015 Apr;45(4):593-605. doi: 10.1007/s00247-014-3210-y. Epub 2015 Apr 1. PMID 25828359
- [Result] Shiff NJ, Brant R, Guzman J, Cabral DA, Huber AM, Miettunen P, Roth J, Scuccimarri R, Alos N, Atkinson SA, Collet JP, Couch R, Cummings EA, Dent PB, Ellsworth J, Hay J, Houghton K, Jurencak R, Lang B, Larche M, Leblanc C, Rodd C, Saint-Cyr C, Stein R, Stephure D, Taback S, Rauch F, Ward LM; Canadian Steroid-associated Osteoporosis in the Pediatric Population Consortium. Glucocorticoid-related changes in body mass index among children and adolescents with rheumatic diseases. Arthritis Care Res (Hoboken). 2013 Jan;65(1):113-21. doi: 10.1002/acr.21785. PMID 22826190
- [Result] Phan V, Blydt-Hansen T, Feber J, Alos N, Arora S, Atkinson S, Bell L, Clarson C, Couch R, Cummings EA, Filler G, Grant RM, Grimmer J, Hebert D, Lentle B, Ma J, Matzinger M, Midgley J, Pinsk M, Rodd C, Shenouda N, Stein R, Stephure D, Taback S, Williams K, Rauch F, Siminoski K, Ward LM; Canadian STOPP Consortium. Skeletal findings in the first 12 months following initiation of glucocorticoid therapy for pediatric nephrotic syndrome. Osteoporos Int. 2014 Feb;25(2):627-37. doi: 10.1007/s00198-013-2466-7. Epub 2013 Aug 16. PMID 23948876
- [Result] Siminoski K, Lentle B, Matzinger MA, Shenouda N, Ward LM; Canadian STOPP Consortium. Observer agreement in pediatric semiquantitative vertebral fracture diagnosis. Pediatr Radiol. 2014 Apr;44(4):457-66. doi: 10.1007/s00247-013-2837-4. Epub 2013 Dec 10. PMID 24323185